CLINICAL TRIAL: NCT00866944
Title: A Randomized, Open-label, Controlled, Multi-center Phase II Study to Evaluate the Efficacy and Safety of Adecatumumab Alone or Sequentially to FOLFOX Relative to FOLFOX After R0 Resection of Colorectal Liver Metastases
Brief Title: Study of Adecatumumab Relative to FOLFOX After R0 Resection of Colorectal Liver Metastases
Acronym: MT201-204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT201-204
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: Colorectal carcinoma; Liver metastases (only); R0 resection; R0 resection of liver metastases from colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — adecatumumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Adecatumumab alone
  Interventions: Drug: Adecatumumab
- 2 (Experimental): FOLFOX 4 followed by Adecatumumab
  Interventions: Drug: Adecatumumab and FOLFOX
- 3 (Active Comparator): FOLFOX 4 alone
  Interventions: Drug: FOLFOX 4

INTERVENTIONS:
Drug: Adecatumumab — Adecatumumab,6-9mg/kg, every 14 days, 24 cycles
  Other Names: MT201
  Arms: 1
Drug: Adecatumumab and FOLFOX — FOLFOX 4, every 14 days, 12 cycles followed by Adecatumumab, 6-9mg/kg, every 14 days, 12 cycles
  Arms: 2
Drug: FOLFOX 4 — FOLFOX 4, every 14 days, 12 cycles
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effect of adecatumumab alone or following FOLFOX in patients with R0 resected liver metastases from CRC (colorectal carcinoma) and to compare the effect to FOLFOX alone.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed complete resection (R0) of liver metastases from colorectal adenocarcinoma
* Age ≥18 years
* ECOG performance status ≤ 2
* Patient was informed, has read and understood the patient information / informed consent form and has given written informed consent

Exclusion Criteria:

* Extra-hepatic distant metastases or locally recurrent disease at time of enrolment
* Neoadjuvant chemotherapy of liver metastases prior to surgery
* Any anticancer chemotherapy within 4 weeks prior to study entry
* Start of Oxaliplatin-based chemotherapy within 9 months prior to study entry
* Any biological anticancer therapy or immunotherapy within 4 weeks prior to study entry
* Any radiotherapy or radio frequency ablation (RFA) to the liver prior to surgery
* Treatment with any investigational product within a time range of 4-5 half-lives (t½) prior to study entry
* Acute or chronic pancreatitis or history of alcohol induced pancreatitis
* Liver cirrhosis, acute hepatitis or chronic hepatic disease
* Any unresolved complications from prior surgery
* Persistent neuropathy
* History of other malignancy within 5 years prior to study start, with the exception of basal cell carcinoma of the skin, carcinoma in situ of the cervix and Ductal Carcinoma in Situ (DCIS)
* History of inflammatory bowel disease
* Active severe infection, any other concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator
* Use of immune-suppressive agents such as the regular use of systemic corticosteroids
* HIV positivity
* Known hypersensitivity or intolerability to immunoglobulins in general, other recombinant human or humanized antibodies, Folinic Acid, 5-Fluorouracil, Oxaliplatin or a component of the study drug formulations, known dihydropyrimidine dehydrogenase (DPD) deficiency
* Pregnant or nursing women
* Women of childbearing potential or male patients not willing to use an effective form of contraception during treatment phase of the study and at least 6 months thereafter
* Not willing or incapable to comply with all study visits and assessments
* Placed into an institution due to juridical or regulatory ruling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Disease free survival rate (DFS) | 1 year

SECONDARY OUTCOMES:
time to relapse | 1 year
Incidence of AEs | 1 year
Quality of Life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Neuhaus, Prof. Dr., Principal Investigator — Charité Campus Virchow Klinikum, Berlin; Patrick Dufour, Pr. Dr., Principal Investigator — Centre Paul Strauss, Strasbourg
Locations (16):
- Centre Paul Strauss, Strasbourg, France
- Germany (15):
  - Zentralklinikum Augsburg, Augsburg
  - Klinikum am Bruderwald, Sozialstiftung Bamberg, Bamberg
  - Charité Campus Virchow Klinikum, Berlin
  - Klinikum der Heinrich-Heine Universität, Düsseldorf
  - J.W. Goethe-Universität, Frankfurt
  - Martin-Luther Universität, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Klinikum der Johannes-Gutenberg Universität, Mainz
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Universitätsklinikum der LMU Grosshadern, München
  - Städtisches Klinikum Neuperlach, München
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum der Universität Regensburg, Regensburg